CLINICAL TRIAL: NCT01379742
Title: Comparison of Health Related Quality of Life and Other Clinical Parameters Between ThinSeed™ and OncoSeed™ for Permanent Low Dose Rate Implantation in Localized Prostate Cancer
Brief Title: Comparison of Between ThinSeed™ and OncoSeed™ for Permanent Prostate Brachytherapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prostate Cancer Foundation of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Thin-1
Record Dates: First submitted 2011-06-20; First posted 2011-06-23 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; prostate brachytherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Needles

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Iodine-125 standard 18 g needle (Active Comparator): Rapidstrand
  Interventions: Device: RapidStrand seeds for use with 18g needle; Device: ThinStrand
- 20 g needle (Active Comparator): Thin Strand
  Interventions: Device: RapidStrand seeds for use with 18g needle; Device: ThinStrand

INTERVENTIONS:
Device: RapidStrand seeds for use with 18g needle — Rapidstrand seeds are standard size and are used with 20 g needles
  Other Names: Both Rapidstrand and Thinstrand are manufactured by Oncura
Device: ThinStrand — ThinStrand seeds are smaller in diameter and used with 20g needles
  Other Names: Both ThinStrand and RapidStrand are manufactured by Oncura.

SUMMARY:
This study will investigate health related quality of life factors in patients undergoing low dose rate prostate brachytherapy. Patients will be randomized to Iodine-125 Thinstrand (for use with 20 g needles) or Rapidstrand (for use with standard 18 g needles). Urinary, bowel, sexual function and bother will be measured by the EPIC questionnaire at various time intervals.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate, clinical stage T1c - T2b, N0, M0
* Greater than or equal to 40 years of age
* Low and Low- Intermediate Risk prostate cancer
* Prostate volumes by TRUS ≤ 60 cc
* I-PSS score < 25 (alpha blockers allowed)
* Signed study-specific informed consent form prior to study entry

Exclusion Criteria:

* Lymph node involvement (N1)
* Evidence of distant metastases (M1)
* Radical surgery for carcinoma of the prostate
* Prior pelvic radiation
* Major medical or psychiatric illness, which in the investigator's opinion would prevent completion of treatment and would interfere with follow- up or ability to complete questionnaires
* Hip prosthesis
* Inability or refusal to provide informed consent
* Evidence of Previous TURP
* Prior hormone therapy
* Prior TURP

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2010-04; Primary Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Health related quality of life including urinary, bowel and sexual function as measured by the EPIC questionnaire | 1 year
  Randomized

CONTACTS AND LOCATIONS:
Overall Officials: Brian J Moran, MD, Principal Investigator — Chicago Prostate Center
Locations (1):
- Chicago Prostate Center, Westmont, Illinois, United States